CLINICAL TRIAL: NCT00306696
Title: A Randomised Study Examining the Effect of Different Diuretics on Fluid Balance in Diabetics Treated With Avandia
Brief Title: Examining the Effect of Different Diuretics on Fluid Retention in Diabetics Treated With Rosiglitazone.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49653/342
Record Dates: First submitted 2006-03-22; First posted 2006-03-24 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus
Keywords: rosiglitazone; fluid retention; Type 2 diabetes; diuretics
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Rosiglitazone; Spironolactone; Hydrochlorothiazide; Furosemide

INTERVENTIONS:
Drug: Rosiglitazone
Drug: spironolactone
Drug: hydrochlorothiazide
Drug: frusemide
  Other Names: spironolactone; hydrochlorothiazide; Rosiglitazone

SUMMARY:
Study examining the effect of different diuretics on fluid retention in diabetics treated with rosiglitazone.

DETAILED DESCRIPTION:
A randomised, open-label, parallel group study to evaluate the management of rosiglitazone-related fluid retention by investigating the effect of diuretics on plasma volume in subjects with type 2 diabetes mellitus treated for twelve weeks with rosiglitazone 4mg bd in addition to background anti-diabetic agents.

ELIGIBILITY:
Inclusion criteria:

* Subjects with type 2 diabetes.
* Stable FPG of >=7.0 and <=12.0mmol/L.
* Subjects had to have been established on SU treatment or SU+MET treatment for at least 2 months.
* Serum creatinine level > 130 micromol/L.

Exclusion criteria:

* Subjects taking > 2 concomitant oral anti-diabetic agents.
* Subjects with HbA1c >=10%.
* Subjects already receiving diuretic medication.
* Subjects unstable or severe angina.
* CHF NYHA class i-iv.
* Subjects with clinically significant hepatic disease.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2002-10; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Changes in Haematocrit following 7 days diuretic adminstration.

SECONDARY OUTCOMES:
Total body fluid & extracellular fluid, body weight, haematocrit & haemoglobin.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (42):
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Sint-Gillis-Waas
- GSK Investigational Site, Winnipeg, Manitoba, Canada
- Denmark (3):
  - GSK Investigational Site, Aarhus
  - GSK Investigational Site, Hellerup
  - GSK Investigational Site, Hvidovre
- France (2):
  - GSK Investigational Site, Dommartin-lès-Toul
  - GSK Investigational Site, Paris
- Germany (6):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Neuss, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Blieskastel, Saarland
  - GSK Investigational Site, Dresden, Saxony
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, N. Efkarpia, Thessaloniki
  - GSK Investigational Site, Nikaia Piraeus
- GSK Investigational Site, Jerusalem, Israel
- Italy (5):
  - GSK Investigational Site, Acquavive Delle Fonti (BA), Apulia
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Perugia, Umbria
- GSK Investigational Site, Utrecht, Netherlands
- Norway (3):
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Stavanger
  - GSK Investigational Site, Tromsø
- Poland (5):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Warsaw
- Slovakia (3):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Ľubochňa
- Spain (4):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Tarrasa, Barcelona
- United Kingdom (3):
  - GSK Investigational Site, Newcastle upon Tyne, Northumberland
  - GSK Investigational Site, Rugby, Warwickshire
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Karalliedde J. Abstract (oral presentation). Management of Rosiglitazone Related Fluid Retention. Diabetes 2005; Vol 54, (suppl 1):Abstract number 81-OR
- [Result] Karalliedde J, Buckingham R, Starkie M, Lorand D, Stewart M, Viberti G; Rosiglitazone Fluid Retention Study Group. Effect of various diuretic treatments on rosiglitazone-induced fluid retention. J Am Soc Nephrol. 2006 Dec;17(12):3482-90. doi: 10.1681/ASN.2006060606. Epub 2006 Nov 8. PMID 17093067
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 49653/342 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 49653/342 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 49653/342 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 49653/342 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 49653/342 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 49653/342 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 49653/342 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register